CLINICAL TRIAL: NCT05242250
Title: A Multi-Center, Real-World Evidence Registry to Assess Outcomes for the Long-Term Impact of Catheter Ablation for Atrial Fibrillation: DYNAMIC AF Registry
Brief Title: Real-World Evidence Registry to Assess Outcomes of Catheter Ablation for Atrial Fibrillation (DYNAMIC AF Registry)
Status: Terminated | Type: Observational
Why Stopped: Decision made to close enrollment in October and close the registry by December 2023
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: DYNAMIC AF
Record Dates: First submitted 2022-01-12; First posted 2022-02-16 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation; atrial fibrillation ablation; catheter ablation; persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Acute SOC Sites with Patients with paroxysmal or persistent atrial fibrillation: Patients with symptomatic, refractory or intolerant to at least one Class I or III AAD, paroxysmal atrial fibrillation (AF episode terminating spontaneously within 7 days) or symptomatic, refractory or intolerant to at least one Class I or III AAD, persistent AF (continuous AF sustained beyond 7-days and less than 1-year) who, in the opinion of the investigator, are candidates for ablation for AF.
  Interventions: Device: Catheter Ablation
- Symptomatic Monitoring SOC Sites with Patients with paroxysmal or persistent atrial fibrillation: Patients with symptomatic, refractory or intolerant to at least one Class I or III AAD, paroxysmal atrial fibrillation (AF episode terminating spontaneously within 7 days) or symptomatic, refractory or intolerant to at least one Class I or III AAD, persistent AF (continuous AF sustained beyond 7-days and less than 1-year) who, in the opinion of the investigator, are candidates for ablation for AF.
  Interventions: Device: Catheter Ablation
- Full Monitoring SOC Sites with Patients with paroxysmal or persistent atrial fibrillation: Patients with symptomatic, refractory or intolerant to at least one Class I or III AAD, paroxysmal atrial fibrillation (AF episode terminating spontaneously within 7 days) or symptomatic, refractory or intolerant to at least one Class I or III AAD, persistent AF (continuous AF sustained beyond 7-days and less than 1-year) who, in the opinion of the investigator, are candidates for ablation for AF.
  Interventions: Device: Catheter Ablation

INTERVENTIONS:
Device: Catheter Ablation — Ablation RF technologies manufactured by Abbott.
  Other Names: Atrial Fibrillation Ablation

SUMMARY:
DYNAMIC AF is an observational, prospective, multi-center, non-randomized registry designed to obtain real world clinical experience of radiofrequency (RF) ablation for the treatment of paroxysmal (PAF) and persistent (PsAF) atrial fibrillation ablation. Patient assessments will occur at pre- procedure, procedure, 12 weeks, 6 months and 1 year post ablation.

DETAILED DESCRIPTION:
Dynamic AF is a prospective, observational, multi-center, non-randomized registry designed to obtain real world clinical experience associated with the use of Abbott technologies for AF ablation. Future technologies may be included as they become available in the market. The registry population will include patients with symptomatic PAF or PsAF that meet all eligibility criteria, who, in the opinion of the investigator, are candidates for AF ablation.

All patients will be treated with commercially approved catheters and the ablation procedure will be conducted based on the current standard of care. Participation in the registry does not influence treatment decisions. All consecutive patients presenting at the institution considered for an RF ablation procedure for symptomatic PAF or PsAF should be screened by the investigator or designated member of the research team for study eligibility

The primary purpose of this registry is to assess procedural efficiencies as well as long term procedural safety and effectiveness of RF ablation in the treatment of patients with paroxysmal or persistent atrial fibrillation. The registry will utilize real world clinical data obtained from the use of commercially available technologies under the authority of a health care practitioner within a legitimate practitioner-patient relationship.

To support the objective of the registry, both patient information and procedure data will be collected. Patient-related data will be collected at a pre ablation office visit, a 12-week post ablation office visit, interim arrhythmia recurrence monitoring at 6- and 12-month post ablation and a 12-month post ablation office visit. Procedure related data collection will include procedural workflow and acute, mid and late onset procedure or device related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic, refractory or intolerant to at least one Class I or III AAD, paroxysmal atrial fibrillation (AF episode terminating spontaneously within 7 days) or symptomatic, refractory or intolerant to at least one Class I or III AAD, persistent AF (continuous AF sustained beyond 7-days and less than 1-year) who, in the opinion of the investigator, are candidates for ablation for AF. Refusal to take AADs for any reason is considered intolerant for the purposes of this protocol.
* Plans to undergo an RF catheter ablation procedure using an ablation catheter manufactured by Abbott
* De Novo ablation unless it is a repeat procedure for a subject whose index procedure is also included in the registry
* 18 years of age or older
* Able and willing to participate in baseline and follow up evaluations for the full length of the registry

Exclusion Criteria:

* Pregnant women
* Individual who cannot read or write, or those who cannot legally consent for themselves
* Participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this registry.
* Long-standing persistent AF (continuous AF sustained >=1 year)
* Previous left atrial surgery for atrial fibrillation
* Having a repeat ablation, unless the subject's index ablation procedure is also included in the registry
* In the opinion of the investigator, any known contraindication to an ablation procedure or to any device or drug required for use during an ablation procedure as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at participating sites for atrial fibrillation ablation that meet all inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Long term safety | 12 months
  Long term safety is assessed by collection of procedure or device related complications.
Long term effectiveness (paroxysmal) | 12 months
  Freedom from atrial arrhythmias (atrial fibrillation/atrial flutter/atrial tachycardia) recurrence (documented episodes greater than 30 seconds) at 12-month follow-up.
Long term effectiveness (persistent) | 12 months
  Freedom from symptomatic atrial arrhythmia (atrial fibrillation/atrial flutter/atrial tachycardia) recurrence (documented episodes greater than 30 seconds) at 12-month follow-up
Procedural efficiency | Immediately after procedure
  Procedure time, ablation time, fluoroscopy time

SECONDARY OUTCOMES:
Acute success | Immediately after procedure
  Termination of clinical arrhythmia, defined by termination to sinus rhythm or non-inducibility of clinical arrhythmia after ablation (cardioversion allowed prior to inducibility attempt)
Patient-reported Outcome | 12 months
  Assessed with 3 items-- How do you feel now compared to pre-ablation: 1) at rest; 2) during mild exercise; and 3) during rigorous exercise
Acute safety | 7 days
  Assessed by collection of procedure or device related complications that occur within 7 days of the ablation procedure
Acute safety | 30 days
  Assessed by collection of peri-procedural complications that occur greater than 7 days but within 30 days post ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Osorio, MD, Principal Investigator — Grandview Medical Center; Paul Zei, PhD, MD, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Grandview Medical Center, Birmingham, Alabama
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Penn Presbyterian Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No